CLINICAL TRIAL: NCT02142946
Title: Quantified Balance Measures During Stance and Gait: Clinical Relevance for Multiple Sclerosis Patients in Comparison to Patients With Inner Ear Balance Problems. A Longitudinal Clinical Study.
Brief Title: Quantified Balance Measures During Stance and Gait: Multiple Sclerosis Patients. A Longitudinal Clinical Study
Acronym: MS-Gait
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-026
Record Dates: First submitted 2014-05-16; First posted 2014-05-20 (Estimated); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Balance Control

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (10):
- RIS MS patients: Radiologically Isolated Syndrome (RIS) MS patients
- CIS MS patients: Clinically Isolated Syndrome (CIS) patients during a stable phase
- RRMS patients: Relapsing-remitting (RR) MS patients during a stable phase
- SPMS Patients: Secondary progressive MS patients (SPMS)
- PPMS Patients: Primary progressive MS patients (PPMS)
- Controls: Age and gender matched controls
- CI Patients: Cochlear Implant patients pre- and post-operatively
- UVL Patients: Unilateral vestibular loss patients in acute and compensated state
- Chronic UVL: Chronic unilateral vestibular loss patients
- Phobic: Phobic vertigo patients

SUMMARY:
The primary objective of this project is to track changes over time in balance control parameters measured during stance and gait for different groups of multiple sclerosis (MS) patients. Our primary goal is to determine whether these changes in balance control over time predict transitions in MS progression to a more disease affected state, and are different from changes over time for patients with balance deficits due to vestibular sensory disorders. A part of this goal is also to determine whether these changes in balance control are correlated with changes in patients' self-reported deficits and are similar to those changes in balance control of patients with peripheral vestibular loss. The secondary objective is to determine for multiple sclerosis (MS) patients the relationship of their balance parameters to different gait speeds, in order to advise them on, and promote via feedback, safe walking speeds. Fulfilling the first of our objectives would lead to better tracking of MS disease changes over time, earlier quantification of onset of symptoms suggesting a worsening of disease status, and, we assume, greater patient satisfaction knowing that quantification of symptoms fits subjective feelings of balance deficits during stance and gait. Achieving the second objective would lead to improved balance during gait. We aim to carry out these objectives using equipment (SwayStar) which we have proven is sensitive to MS induced balance deficits {2}, but costs far less to operate and maintain than previously used quantification tools. We aim to investigate the balance deficits during gait in different MS patient groups using a multimodal approach with a SwayStar system (analysis of balance during stance and gait in terms of trunk-pelvis movements near the centre of mass) and patient questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Balance deficits due to inner ear disease or MS

Exclusion Criteria:

* Inability to walk without a walking aid

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with MS or UVL
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in balance during stance and gait | 1 year
  Measurement of trunk sway as balance measure during stance and gait trials

CONTACTS AND LOCATIONS:
Overall Officials: John HJ Allum, DSc, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Lab for Exp Otoneurology, University Hospital Basel, Basel, Switzerland